CLINICAL TRIAL: NCT01355900
Title: Influence of the Intraoperative Tourniquet Application Method on the Perioperative Blood Loss, Frequency of Transfusion and Close Postoperative Outcomes in Primary Total Knee Arthroplasty Patients
Brief Title: Comparison of Three Tourniquet Application Methods in Primary Total Knee Arthroplasty Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Narunas Porvaneckas, Pofessor, PhD, Vilnius University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP-001
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Knee Osteoarthritis
Keywords: Total knee arthroplasty; Tourniquet; Blood loss; Volume loading test
MeSH Terms: conditions — Osteoarthritis, Knee; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- I tourniquet tactic (Other): Use volume loading test twice (before surgery and 24hrs postoperatively). Total knee arthroplasty performed under tourniquet. Lower limb tourniquet inflation- before incision, deflation- after bone cement set.
  Interventions: Procedure: Total knee arthroplasty performed under tourniquet
- II tourniquet tactic (Other): Use volume loading test twice (before surgery and 24hrs postoperatively). Total knee arthroplasty performed under tourniquet. Lower limb tourniquet inflation- before cement application, deflation- after bone cement set.
  Interventions: Procedure: Total knee arthroplasty performed under tourniquet
- III tourniquet tactic (Other): Use volume loading test twice (before surgery and 24hrs postoperatively). Total knee arthroplasty performed under tourniquet. Lower limb tourniquet inflation- before incision, deflation- after wound closure
  Interventions: Procedure: Total knee arthroplasty performed under tourniquet
- IV control group (Other): Do not use volume loading test. Total knee arthroplasty performed under tourniquet. Lower limb tourniquet inflation- before cement application, deflation- after bone cement set.
  Interventions: Procedure: Total knee arthroplasty performed under tourniquet

INTERVENTIONS:
Procedure: Total knee arthroplasty performed under tourniquet — Comparison of the different tourniquet tactics.
  Other Names: Volume loading test

SUMMARY:
Different strategies of tourniquet application during elective primary total knee arthroplasty are thought to be associated with different outcomes. In that context, the study investigates different tactics in the search of optimal application of the tourniquet and the related fluid management during 24 perioperative hours.

DETAILED DESCRIPTION:
The optimal application of tourniquet should reduce perioperative blood loss, create bloodless operative field, improve cementing technique and shorten surgery time. Meanwhile, inadequate application may increase the risk of deep vein thrombosis and pulmonary thromboembolism. Previous attempts to compare the tourniquet strategies in respect to the perioperative blood loss did not show significant difference. The investigators use the volume loading test aiming to optimize the fluid status and obtain the hemoglobin concentration in the conditions of standardized plasma dilution. The test is deployed just before the surgery and after postoperative 24 hrs in ICU. Functional outcomes and possible length of hospital stay is also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis of the knee undergoing total knee arthroplasty with spinal-epidural anesthesia
* Age > 50 and < 80 years
* ASA (American Society of Anesthesiology Classification) II physical status
* Signed informed consent form

Exclusion Criteria:

* History of a bleeding disorder
* Current chronic anticoagulation therapy
* History of DVT (Deep Vein Thrombosis), thromboembolic complications, acute cardiac insufficiency
* Anemia before surgery required blood transfusion
* ASA I, ASA>=III physical status
* Age < 50 and > 80 years
* BMI (Body Mass Index) < 20 and > 40kg/m2
* Intravascular fluid infusion within 24 hours before study
* Chronic non-steroidal anti-inflammatory drug use (more than 6month daily use)
* Rheumatoid arthritis
* Diabetes mellitus
* Psychiatric illness (intake of other psychiatric medication than selective serotonin reuptake inhibitors)
* Alcohol intake 5 U daily
* Contraindication to epidural catheter insertion
* Surgery not by project surgeon
* Participation in the other study
* Active malignancy
* Previous open knee surgery

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Perioperative blood loss. | Before (baseline) the surgery and 24 hrs postoperatively
  The volume loading test is deployed for the comparison of perioperative hemoglobin in the standardized plasma dilution.

SECONDARY OUTCOMES:
Wound healing | Within 6 days postoperatively
Hemodilution | Within 6 days postoperatively
Cardiac stroke volume | Within 6 days postoperatively
Body temperature | Within 6 days postoperatively
Pain (Visual Analog Scale) | Within 6 days postoperatively
Number of opiate injections | Within 6 days postoperatively
Straight-leg raising test | Within 6 days postoperatively
Timed up and go test | Within 6 days postoperatively
Knee flexion, extension, extension lag | Within 6 days postoperatively
Knee swelling | Within 6 days postoperatively
Complications | Within 6 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Narunas Porvaneckas, PhD, Principal Investigator — Medical Faculty of Vilnius University, Clinic of Rheumatology, Traumatology and reconstructive surgery
Locations (1):
- Republic Vilnius University Hospital, Vilnius, Lithuania

REFERENCES:
- [Result] Kvederas G, Porvaneckas N, Andrijauskas A, Svensen CH, Ivaskevicius J, Mazunaitis J, Marmaite U, Andrijauskas P. A randomized double-blind clinical trial of tourniquet application strategies for total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2013 Dec;21(12):2790-9. doi: 10.1007/s00167-012-2221-1. Epub 2012 Sep 28. PMID 23052115